CLINICAL TRIAL: NCT01665729
Title: Diagnosis and Treatment of Minor Ischaemic Stroke According to the Etiology and Pathogenesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Li Haiyan (Other)
Responsible Party: Sponsor-Investigator, Li Haiyan, Dr., Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: 2011-2-48
Record Dates: First submitted 2012-08-12; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Ischaemic Stroke
Keywords: etiology; pathogenesis; minor ischaemic stroke; types; intervention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- artery-artery embolus: There is no hypoperfusion ( contralateral compensatory is good )
- Hypoperfusion: Contralateral compensatory not sufficient
- Hypoperfusion and embolus amotic: Hypoperfusion and embolus amotic

SUMMARY:
Negligence or contempt of the etiology and pathogenesis of minor ischaemic stroke in the early diagnosis and effective treatment leads to more than 40-50% of patient with recurrent episodes, and 10% patient died. Therefore, diagnosis and treatment of minor ischaemic stroke according to the etiology and pathogenesis is important.

The 2007 Korean modified TOAST type got some progress, but there exists two major disadvantages: imperfect diagnosis and pathogenesis of perforator artery infarction etiology; lack of typing according to the pathogenesis of large atherosclerotic infarction and taking measures of treatment according to the new types. Recently, domestic professor Gaoshan proposes new approach to diagnose and treat minor ischaemic stroke according to the etiology and pathogenesis of CISS typing, but the pathogenesis of hypoperfusion infarction with severe stenosis of large artery is unclear. Is it low perfusion? Or artery-artery embolization? Or both? How to distinguish the pathogenesis of branch artery disease: by atherosclerosis? Or hyalinosis? Or both? How to check the validity of clinical types? This study take different interventions according to different types and observation of the long term clinical results of intervention( mortality, recurrence rate, disability rate and rate of cerebral hemorrhage and subarachnoid hemorrhage), in order to clarify the new types can indeed solve the current problem of minor ischaemic stroke with high mortality, recurrence rate, disability rate and rate of cerebral hemorrhage and subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

one of two conditions:

1. conscious patients with any of NIHSS score = 1,or
2. NIHSS ≤ 3

Exclusion Criteria:

* patients Over 80 years of age
* patients With serious heart, lung, liver, kidney dysfunction or
* severe systemic complications,
* a known tumor,
* pregnancy,
* having a history of cerebral hemorrhage

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with new emergence of minor ischaemic stroke ( one of two conditions: (1) conscious patients with any of NIHSS score = 1,or (2) NIHSS ≤ 3 )
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zhengqi Lu, prof., Study Chair — Department of Neurology,The Third Afﬁliated Hospital of Sun yat-sen University
Locations (1):
- Department of Neurology,The Third Afﬁliated Hospital of Sun yat-sen University, Guangzhou, Guangdong, China